CLINICAL TRIAL: NCT01832051
Title: HER2-PET as a Diagnostic Tool in Breast Cancer Patients With a Clinical Dilemma
Brief Title: Clinical Value of 89Zr-trastuzumab PET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, C.P. Schroder, MD, PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Her2.4
Record Dates: First submitted 2013-04-03; First posted 2013-04-15 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2-PET; 89Zr-trastuzumab; metastatic breast cancer; clinical dilemma
MeSH Terms: conditions — Breast Neoplasms | interventions — zirconium-89-trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HER2-PET (Experimental): Injection of 89Zr-trastuzumab followed by PET scan
  Interventions: Drug: 89Zr-trastuzumab injection

INTERVENTIONS:
Drug: 89Zr-trastuzumab injection

SUMMARY:
Information about the presence of human epidermal growth factor receptor 2 (HER2) in tumor lesions in breast cancer patients is essential for diagnostic and therapeutic management of metastatic breast cancer. In daily practice however, obtaining a metastasis biopsy can be difficult or impracticable. Therefore, clinicians can be faced with a persistent clinical dilemma in some breast cancer patients, leading to suboptimal therapy decisions due to lack of HER2 receptor information. Circulating tumor cells (CTCs), which may provide additional information, have so far not been able to replace the biopsy. To solve this problem, non-invasive whole body visualization and quantification of HER2 expression by means of the HER2-PET may be a valuable tool.

In this prospective multicenter imaging study, eligible patients will receive one HER2-PET and CTC analysis in addition to standard work up for metastatic disease. Subsequent administration of anti-HER2 therapy will be evaluated. Referring physicians fill in three questionnaires, one before HER2-PET and two after HER2-PET.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a history of histological and/or cytological proven HER2-positive primary breast cancer. In the Netherlands HER2-positivity is defined as:

   * HER2 immunohistochemical score of 3+, or
   * HER2 immunohistochemical score of 2+ and positive FISH for HER2/c-erbB2 amplification.

   In Belgium HER2-positivity is defined as positive FISH for HER2/c-erbB2 amplification.
2. Patients with suspected metastatic disease or local recurrence of HER2-positive breast cancer and a clinical dilemma:

   * in whom standard work up with imaging has failed to solve the clinical dilemma (diagnostic/therapeutic), leaving issues with regard to HER2 status of lesions and
   * in whom a biopsy is desirable but cannot (easily) be performed due to technical or patient factors or otherwise.
3. Standard work-up with imaging is defined as CT chest and abdomen, bone scintigraphy, as well as FDG-PET.
4. Age >18 years of age.
5. WHO performance status 0-2.
6. Signed written informed consent.
7. Able to comply with the protocol.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Prior allergic reaction to immunoglobulins or immunoglobulin allergy.
3. Inability to comply with study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Concordance between HER2-PET results and anti-HER2 therapy | about 2 years (end of study)
  Concordance between HER2-PET results and anti-HER2 therapy is defined as HER2 positive lesion(s) on HER2-PET and subsequent anti-HER2 therapy; or no HER2 positive lesions on HER2-PET and no subsequent anti-HER2 therapy. It is considered a clinically relevant contribution of HER2-PET to anti-HER2-therapy decisions if there is a concordance in at least 2/3 of included patients.

SECONDARY OUTCOMES:
Correlation of HER2-PET results and questionnaire results regarding clinical value of HER2-PET for the referring clinician | about 2 years (end of study)
  Correlation of HER2-PET result (assessed about 1 week after scan) and questionnaire results (before, directly after, and 3 months after scan)
Correlation of HER2-PET results with standard conventional work-up | about 2 years (end of study)
  Correlation of HER2-PET result (assessed about 1 week after scan) and standard conventional work-up (assessed before/at screening)
Correlation of HER2-PET results and HER-2 expression by CTCs | about 2 years (end of study)
  Correlation of HER2-PET result (assessed about 1 week after scan) and HER-2 expression by CTCs (blood for CTC analysis will be drawn at day of tracer injection, analysis within 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: C.P. Schröder, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center, Groningen, Netherlands